CLINICAL TRIAL: NCT06788899
Title: Clinical Audit on Uterine Closure During Caesarean Section in Assiut Women's Health Hospital
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Lobna Hassan Ahmed AbdelRhman, Principal investigator, Assiut University
Other Study IDs: Uterus closure
Record Dates: First submitted 2024-12-22; First posted 2025-01-23 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2024-12

CONDITIONS: Uterine Closure in Caesarean Section

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Auditing of closure of uterine incision in Caesarean section in Assiut Women's Health Hospital.

ELIGIBILITY:
Inclusion Criteria:

* all elective Caesarean section

Exclusion Criteria:

1. Placenta previa
2. Chorioamionitis
3. PROM
4. Diabetic women
5. Immunocompromised women
6. Women with heart disease
7. Women with renal or liver disease
8. Women on corticosteroids therapy
9. Preeclampsia
10. Women with hypertensive disorders

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All elective Caeserean sections with no medical or obestetric disorder
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Improve performance of closure of Caesarean section. in Assiut Women health hospital according to NICE guidelines and National Library of Medicine | Through study completion an average of one year
  Questionaire

SECONDARY OUTCOMES:
Decrease complications of caeserean section | Through study completion an average of one year
  Questionaire
Training of university staff | Through study completion an average of one year
  Questionaire

REFERENCES:
- [Background] Principles of Methodological Design of Clinical Audit. Arch Med Vol No:10 Iss No:2:2(1)
- [Background] 1-Morrell C and Harvey G (1999) The Clinical Audit Handbook. Improving the quality of health care. London: Bailliere Tindall.(1)
- [Background] Hauth JC, Owen J, Davis RO. Transverse uterine incision closure: one versus two layers. Am J Obstet Gynecol. 1992 Oct;167(4 Pt 1):1108-11. doi: 10.1016/s0002-9378(12)80048-2. PMID 1415400